CLINICAL TRIAL: NCT05755620
Title: A Phase 1, Open-Label, Comparator-Controlled, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of a Single Dose of VRC H1ssF-3928 mRNA-LNP in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Immunogenicity of a Single Dose of H1ssF-3928 mRNA-LNP in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 21-0010; 75N93019C00054
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2023-06-23

CONDITIONS: Influenza
Keywords: Comparator-Controlled; Dose-Escalation; H1ssF-3928; Healthy Adults; mRNA-LNP; Phase 1
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1, Low Dose (Experimental): 10 healthy adult volunteer subjects from 18-49 years of age are split into two subgroups. The sentinel subgroup includes 2 vaccine recipients who will receive 10 mcg of the H1ssF_3928 mRNA Vaccine, administered intramuscularly once. The sentinel subgroup is observed for 8 days to monitor any early vaccine related adverse events. After the observation period, the remaining participants will receive the same dosage, 10 mcg of the H1ssF 3928 mRNA vaccine administered intramuscularly once. N = 10
  Interventions: Other: Sodium Chloride, 0.9%; Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Arm 2, Medium Dose (Experimental): 10 healthy adult volunteer subjects from 18-49 years of age are split into two subgroups. The sentinel subgroup includes 2 vaccine recipients who will receive 25 mcg of the H1ssF_3928 mRNA Vaccine, administered intramuscularly once. The sentinel subgroup is observed for 8 days to monitor any early vaccine related adverse events. After the observation period, the remaining participants will receive the same dosage, 25 mcg of the H1ssF 3928 mRNA vaccine administered intramuscularly once. N = 10
  Interventions: Other: Sodium Chloride, 0.9%; Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Arm 3, High Dose (Experimental): 10 healthy adult volunteer subjects from 18-49 years of age are split into two subgroups. The sentinel subgroup includes 2 vaccine recipients who will receive 50 mcg of the H1ssF_3928 mRNA Vaccine, administered intramuscularly once. The sentinel subgroup is observed for 8 days to monitor any early vaccine related adverse events. After the observation period, the remaining participants will receive the same dosage, 50 mcg of the H1ssF 3928 mRNA vaccine administered intramuscularly once. N = 10
  Interventions: Other: Sodium Chloride, 0.9%; Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Arm 4, Optimal Dose (Experimental): 10 healthy adult volunteer subjects from 18-49 years of age will receive the selected optimal dose of the H1ssF_3928 mRNA Vaccine, administered intramuscularly once. The optimal dosing group will be selected based on safety outcomes from the 10 mcg, 25 mcg, and 50 mcg dosing groups. For the optimal dose, the highest dose with no identified safety concerns as determined by the Safety Review Committee (SRC) will be selected. N =10
  Interventions: Other: Sodium Chloride, 0.9%; Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Arm 5, IIV4 (Active Comparator): 10 healthy adult volunteer subjects from 18-49 years of age will receive licensed Quadrivalent Influenza Vaccine (IIV4), administered intramuscularly once. Subjects receiving IIV4 will be followed for safety, but only their immune responses will be compared to those of participants receiving H1ssF_3928 mRNA Vaccine. N=10
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine

INTERVENTIONS:
Biological: Influenza Virus Quadrivalent Inactivated Vaccine — A seasonal quadrivalent inactivated influenza vaccine (IIV4), prepared from influenza viruses propagated in embryonated chicken eggs, protecting against 2 influenza A subtypes and 2 influenza B subtypes.
  Arms: Arm 5, IIV4
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection
  Arms: Arm 1, Low Dose; Arm 2, Medium Dose; Arm 3, High Dose; Arm 4, Optimal Dose
Biological: VRC-FLUNPF099-00-VP (H1ssF_3928) — The vaccine consists of modified nucleoside messenger RNA (mRNA) encapsulated in lipid nanoparticles (LNP), comprised of four lipid components: (ALC-307 (ionizable lipid), DSPC, cholesterol, and ALC-0159 [PEG lipid]).
  Arms: Arm 1, Low Dose; Arm 2, Medium Dose; Arm 3, High Dose; Arm 4, Optimal Dose

SUMMARY:
This is a Phase 1, single-site, open-label, comparator-controlled dose escalating study of an intramuscularly (IM) administered mRNA-LNP vaccine encoding for (Vaccine Research Center) VRC H1ssF 3928 of up to 50 healthy adult volunteers aged 18 to 49 years, inclusive. This study is designed to assess the safety and immunogenicity of one dose of H1ssF 3928 mRNA Vaccine. Eligible participants will be sequentially enrolled into dosing groups (10 mcg, 25 mcg, and 50 mcg, selected optimal dose) to receive the H1ssF 3928 mRNA Vaccine at the specified dose. A separate group of 10 participants will receive licensed quadrivalent influenza vaccine (IIV4). Subjects receiving IIV4 will be followed for safety but only their immune responses will be compared to those of participants receiving H1ssF 3928 mRNA Vaccine. Dosing of H1ssF 3928 mRNA Vaccine will commence at the lowest dose (10 mcg) and only escalate to the next highest dose if safety concerns are not identified. Up to ten subjects will be enrolled per dosing cohort. Reactogenicity and adverse event (AE) information through Day 7 and clinical laboratory results through Day 8 from the first three dosing groups will guide the selection of an optimal dose group to include 10 subjects who will receive the optimal dose of mRNA-LNP. The primary objective of this study is to assess the safety of a single dose of VRC H1ssF 3928 mRNA-LNP vaccine administered IM in healthy adults, 18-49 yrs, at doses of 10 mcg, 25 mcg, and 50 mcg.

DETAILED DESCRIPTION:
This is a Phase 1, single-site, open-label, comparator-controlled dose escalating study of an intramuscularly (IM) administered mRNA-LNP vaccine encoding for (Vaccine Research Center) VRC H1ssF 3928 of up to 50 healthy adult volunteers aged 18 to 49 years, inclusive. This study is designed to assess the safety and immunogenicity of one dose of H1ssF 3928 mRNA Vaccine. Eligible participants will be sequentially enrolled into dosing groups (10 mcg, 25 mcg, and 50 mcg, selected optimal dose) to receive the H1ssF 3928 mRNA Vaccine at the specified dose. A separate group of 10 participants will receive licensed quadrivalent influenza vaccine (IIV4). Subjects receiving IIV4 will be followed for safety but only their immune responses will be compared to those of participants receiving H1ssF 3928 mRNA Vaccine. Dosing of H1ssF 3928 mRNA Vaccine will commence at the lowest dose (10 mcg) and only escalate to the next highest dose if safety concerns are not identified. For each VRC H1ssF 3928 mRNA-LNP (Lipid Nanoparticle) dosing group, the first two subjects enrolled will be considered the sentinel subgroup. After the two subjects in the Low Dose sentinel subgroup are enrolled and given their vaccination, enrollment will then be stopped pending a review of the reactogenicity and safety data collected through Day 3 for both subjects. Approval by the reviewing group will allow for continued enrollment of the remaining Low Dose Group subjects to complete enrollment of 10 participants. After Low Dose Group enrollment is completed, enrollment will be stopped pending an Safety Review Committee (SRC) review of the reactogenicity and adverse event (AE) information through Day 7 and clinical laboratory results through Day 8 for all Low Dose Group subjects. Approval will allow dose escalation and initiation of enrollment of the Medium Dose Group sentinel subgroup. After the two subjects in the Medium Dose sentinel subgroup are enrolled and given their vaccination, enrollment will then be stopped pending a safety review of the sentinel subgroup as specified for the Low Dose Group. Approval will allow for continued enrollment of Medium Dose Group subjects to complete enrollment of 10 participants. After the Medium Dose Group enrollment is completed, enrollment will be stopped pending an SRC review of the reactogenicity and adverse event information through Day 7 and clinical laboratory results through Day 8 for all Medium Dose Group subjects. Approval will allow dose escalation and initiation of enrollment of the High Dose Group sentinel subgroup. After the two subjects in the High Dose sentinel subgroup are enrolled and given their vaccination, enrollment will then be stopped pending a safety review of the sentinel subgroup as specified for the Low and Medium Dose Groups. Approval will allow for continued enrollment of High Dose Group subjects to complete enrollment of 10 participants. After the High Dose Group enrollment is completed, enrollment will be stopped pending an SRC review of the reactogenicity and adverse event information through Day 7 visit and clinical laboratory results through Day 8 for all High Dose Group subjects. Reactogenicity and AE information through Day 7 and clinical laboratory results through Day 8 from the first three dosing groups will guide the selection of an optimal dose group to include an additional 10 subjects who will receive the optimal dose of mRNA-LNP. The primary objective of this study is to assess the safety of a single dose of VRC H1ssF 3928 mRNA-LNP vaccine administered IM in healthy adults, 18-49 yrs, at doses of 10 mcg, 25 mcg, and 50 mcg. The secondary objective of this study is to assess serum antibody responses to a single dose of VRC H1ssF 3928 mRNA-LNP vaccine administered IM in healthy adults at doses of 10 mcg, 25 mcg, and 50 mcg in comparison to a standard dose of IIV4.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedure.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant, non-breastfeeding females, 18 to 49 years of age, inclusive at time of screening and enrollment.
4. Must agree to collection of venous blood and nasal absorption specimens per protocol and enrollment in DMID Protocol No. 19-0025 biorepository protocol for secondary research and use of residual biologic specimens.
5. Are in good health* and do not have clinically significant medical, psychiatric, chronic or intermittent health conditions including those listed in Exclusion Criteria (Section 1).

   *As determined by medical history, medication use, and physical examination to evaluate ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would not affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. These medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, emergency room [ER] or urgent care for condition [excluding musculoskeletal conditions], or invasive medical procedure and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose or in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening or treatment of continued symptoms of medical diagnosis or condition. Note: Low dose topical, corticosteroids as outlined in the Subject Exclusion Criteria (see Section 1) as well as herbals, vitamins and supplements are permitted.
6. Does not have an ongoing symptomatic condition* for which subject has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan.

   *e.g., ongoing fatigue without a diagnosis for symptom.
7. Pulse is 50 to 100 beats per minute, inclusive.
8. Systolic blood pressure is 90 to 140 mmHg, inclusive.
9. Diastolic blood pressure is 55 to 90 mmHg, inclusive.
10. Body mass index (BMI) of 18 kilograms/square meter (kg/m^2) (inclusive) to <35 kg/m^2 at screening
11. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least 1 acceptable primary form of contraception.***

    *Not of child bearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, salpingectomy, or Essure placement with history of documented radiological confirmation test at least 90 days after the procedure).

    **True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).
    * Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the study product, tubal ligation, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.
    * Must use at least one acceptable primary form of contraception or true abstinence for at least 30 days prior to receipt of study product and at least one acceptable primary form of contraception or true abstinence for at least 30 days following receipt of study product.
12. Women of childbearing potential must have a negative serum HCG pregnancy test at screening and a negative urine HCG pregnancy test within 24 hours prior to the study vaccination.
13. Male participants receiving VRC H1ssF_3928 mRNA-LNP must agree to refrain from donating sperm and to use contraception until Day 60 after vaccination.*

    * Acceptable contraception includes abstinence from intercourse with a female of childbearing potential or use of a male condom when engaging in any activity that allows for passage of ejaculate to a female during the intervention period for at least 60 days after study vaccination.
    * Males in the immunogenicity comparator group do not have to refrain from sperm donation or abstain from intercourse or agree to use a male condom for purposes of this study.
14. Must have received at least one licensed seasonal influenza vaccine within the previous 5 seasons.

Exclusion Criteria:

1. Have an acute illness* or fever (body temperature > / = 38.0 degrees Celsius/100.4 degrees Fahrenheit), as determined by the site Principal Investigator (PI) or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation.*

   * Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Has a screening laboratory* > Grade 1.

   *White blood cell count, absolute neutrophil count, absolute lymphocyte count, hemoglobin, platelet count, prothrombin time (PT), activated partial thromboplastin time (APTT), fibrinogen, creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin, lipase.
4. Has a positive urine toxicology screen (i.e., non-prescribed amphetamines, cocaine, and opiates).
5. Electrocardiogram (ECG) is deemed to be clinically significant by the PI or appropriate sub-investigator.
6. Total iron binding capacity, iron, ferritin and troponin (hsTnl) outside the laboratory normal range at screening.
7. Have any known or suspected immunosuppressive condition, acquired or congenital, or autoimmune conditions as determined by history and/or physical examination.
8. Have immunosuppression as result of treatment including a recent history (within 6 months prior to administration of study vaccine) or use of immunosuppressive or other immune-modifying drugs.
9. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
10. Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
11. Have known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection at screening.
12. Have a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or HIV types 1 or 2 antibodies at screening.
13. Have known chronic liver disease, including fatty liver disease.
14. Have a known allergy or severe allergic reaction to any components of the study vaccine (including polyethylene glycol [PEG]) or the seasonal influenza vaccine (including egg protein).
15. Have a history of a severe reaction following previous immunization with an investigational, authorized, or approved influenza vaccine or mRNA or LNP-containing vaccine containing vaccine.
16. Have a history of Guillain-Barré Syndrome.
17. Have a known history of myocarditis or pericarditis.
18. Have a history of alcohol or drug abuse within 3 years prior to study vaccination.
19. Have any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere* with subject compliance or safety evaluations.

    *As determined by the site PI or appropriate sub-investigator.
20. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
21. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination. Intranasal or topical (skin or eyes) corticosteroids are permitted.
22. Have taken high-dose inhaled or nebulized corticosteroids* within 30 days prior to study vaccination.

    *High-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE
23. Have any significant disorder of coagulation requiring ongoing or intermittent treatment.
24. Have received seasonal influenza vaccine within 90 days prior to enrollment or plans to receive a seasonal influenza vaccine 60 days after study vaccination.
25. Have received any approved or authorized vaccines other than seasonal influenza vaccine within 60 days before enrollment or plans to receive an approved or authorized vaccine 60 days after study vaccination.
26. Have a known history of documented influenza infection within the past 90 days.
27. Have a history of receipt of an investigational H1 influenza vaccine within the past 10 years.
28. Have a history of receipt of a ferritin-based vaccine or an investigational H5 influenza vaccine.
29. Previous participation in DMID Protocol No. 18-0010 human influenza challenge study.
30. Received immunoglobulin and/or any blood products (except Rho D immunoglobulin) within the 90 days prior to study vaccination.
31. Received an experimental agent *within 60 days prior to the study vaccination or expect to receive another experimental agent during the trial-reporting period.**

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this trial
32. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the trial-reporting period.*

    * Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
    * Approximately 12 months after the first study vaccination.
33. The subject has any abnormality or permanent body art (e.g., tattoo) that, in the opinion of the investigator or appropriate sub-investigator, would obstruct the ability to observe local reactions at the injection site.
34. Donation of blood or blood products within 30 days prior to dosing and plans to donate within 60 days following dosing.
35. Has had significant exposure to someone with laboratory-confirmed severe acute respiratory syndrome (SARS-CoV-2) infection or influenza in the 14 days prior to screening or during the period between screening and enrollment visit.*

    *Defined by the Centers for Disease Control and Prevention (CDC) as a close contact with someone who has COVID-19.
36. Has had a positive SARS-CoV-2 test (home or laboratory-based) within 14 days prior to the screening visit or during the period between screening and enrollment visits.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events of special interest (AESIs) corresponding to myocarditis, pericarditis, or myopericarditis with VRC H1ssF_3928 mRNA-LNP vaccine | Day 1 through Day 57
Occurrence of any adverse events of special interest (AESIs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 366
  adverse events of special interest (AESIs) corresponding to Grade 2 or greater decrease in lymphocyte or neutrophil count
Occurrence of any influenza-like illnesses (ILIs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 366
Occurrence of any new-onset chronic medical conditions (NOCMCs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 366
Occurrence of any serious adverse events (SAEs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 366
Occurrence of any unsolicited adverse events (AEs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 28
Occurrence of clinical laboratory adverse events (AEs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 57
Occurrence of medically attended adverse events (MAAEs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 366
Occurrence of solicited reactogenicity adverse events (AEs) with VRC H1ssF_3928 mRNA-LNP vaccine. | Day 1 through Day 14
  Both local and systemic adverse events will be assessed

SECONDARY OUTCOMES:
Geometric mean fold rise (GMFR) of anti-stalk serum antibodies measured by enzyme linked immunosorbent assay (ELISA). | Day 1 through Day 57
Geometric mean fold rise (GMFR) of homologous H1-specific neutralizing antibodies in a reporter microneutralization assay. | Day 1 through Day 57
Geometric mean fold rise (GMFR) of homologous H1-specific neutralizing antibodies in a viral microneutralization assay. | Day 1 through Day 57
Geometric mean titers (GMT) of homologous H1-specific neutralizing antibodies in a reporter microneutralization assay. | Day 1 through Day 57
Geometric mean titers (GMT) Of homologous H1-specific neutralizing antibodies in a viral microneutralization assay. | Day 1 through Day 57
Geometric mean titers of anti-stalk serum antibodies measured by enzyme linked immunosorbent assay (ELISA). | Day 1 through Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Vaccine and Trials Unit, Durham, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05755620/ICF_000.pdf